CLINICAL TRIAL: NCT06682702
Title: The Effectiveness of Dynamic Neuromuscular Stabilization Breathing Exercises in Addition to Schroth Exercises in Individuals With Adolescent Idiopathic Scoliosis
Brief Title: Effectiveness of Dynamic Neuromuscular Stabilization Breathing Exercises With Schroth in Adolescent Idiopathic Scoliosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, MERVE BAŞARDI, Physiotherapist, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-PT-MRVB-RCT
Record Dates: First submitted 2024-10-22; First posted 2024-11-12 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS)
Keywords: rehabilitation; surgery; therapy; Rehabilitation Exercise; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Model description training and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DNS Group (Experimental): Patients diagnosed with adolescent idiopathic scoliosis participated in sessions twice a week for 8 weeks, with each session lasting 45 minutes. During the sessions, ISST Schroth exercises were combined with dynamic neuromuscular stabilization exercises.
  Interventions: Other: DNS Group
- Schroth Group (Experimental): Patients diagnosed with adolescent idiopathic scoliosis participated in sessions twice a week for 8 weeks, with each session lasting 45 minutes. During the sessions, ISST Schroth exercises were performed.
  Interventions: Other: Schroth Group

INTERVENTIONS:
Other: DNS Group — ISST Schroth exercises are a model of exercise aimed at correcting scoliosis in three dimensions. Dynamic neuromuscular stabilization exercises, on the other hand, are designed to achieve sagittal stabilization by utilizing the stabilizing function of the thoracic diaphragm muscle.
  Other Names: Schroth Exercise; Dynamic Neuromuscular Stabilization
  Arms: DNS Group
Other: Schroth Group — ISST Schroth exercises are a model of exercise aimed at correcting scoliosis in three dimensions.
  Other Names: Schroth Exercise
  Arms: Schroth Group

SUMMARY:
In our study, the degree of scoliosis curvature in volunteers will be determined using full-body standing X-rays. Additionally, the rotation degree of the spinal curvature in volunteers will be assessed with a scoliosis meter (a type of ruler) through the forward bending test while standing. To measure the impact of scoliosis on the quality of life, the SRS-22 questionnaire, consisting of 22 questions, will be used. The level of pain experienced by volunteers as a result of scoliosis will be evaluated using the visual analog scale (VAS), where pain intensity is marked on a 10 centimeter line. Lastly, the volunteers; breathing patterns will be assessed by measuring chest circumference with a tape measure.

DETAILED DESCRIPTION:
In this randomized controlled trial, we aim to assess various physical and quality of life parameters in volunteers with scoliosis. The degree of spinal curvature will be measured using full body standing X-rays, providing a detailed assessment of the scoliosis angle. Additionally, the rotation degree of the spinal curvature will be evaluated with a scoliosis meter during the forward bending test, which is commonly used to gauge the rotational component of scoliosis.

Quality of life will be assessed using the Scoliosis Research Society-22 (SRS-22) questionnaire, a validated tool consisting of 22 questions designed to evaluate function, pain, self image, mental health, and satisfaction in individuals with scoliosis. To quantify pain levels experienced due to scoliosis, the Visual Analog Scale (VAS) will be used, in which participants mark their pain intensity on a 10 centimeter line, ranging from "no pain" to "worst pain imaginable." This provides an accurate, subjective measure of pain severity.

Breathing patterns will also be evaluated by measuring the volunteers' chest circumference at full inspiration and expiration using a standard tape measure, allowing us to assess any potential restrictions in lung expansion related to the spinal curvature. Through this comprehensive evaluation, we hope to gain a clearer understanding of how scoliosis affects both the physical and psychological well being of individuals and identify potential areas for therapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically measured Cobb angle value between 10 degrees and 50 degrees
* Age between 10 and 18
* Being diagnosed with Adolescent Idiopathic Scoliosis by a physician
* Being between 0 and 5 in the radiologically determined Risser sign
* Being between 12-25 kg/m2 according to body mass index measurement

Exclusion Criteria:

* Having had any surgery related to scoliosis
* Having been diagnosed with any psychiatric disease
* Having been diagnosed with an oncological disease
* Having a neurological disease, vestibular or visual problem
* Having any pathology that will affect motor performance
* Using medication that affects the central nervous system
* Having been diagnosed with a rheumatological disease
* Having been diagnosed with any cardiovascular disease

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-03-07 (Estimated)

PRIMARY OUTCOMES:
Cobb Angel | 8 weeks
  The Cobb angle will be measured using standing full-spine X-rays to quantify the degree of spinal curvature in patients with scoliosis.
Respiratory Muscle Strength | 8 weeks
  Respiratory muscle strength was measured using an electronic mouth pressure measuring device (Cosmed Ponyy Fx, Rome, Italy). Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) were measured.
Angle Trunk Rotation | 8 weeks
  The Adams forward bending test, commonly used in scoliosis screening, involves positioning the patient with arms extended forward to assess for asymmetric protrusions and coronal imbalance in the back, while a scoliometer is utilized to measure the degree of spinal rotation and track progression of trunk asymmetry and deformity.

SECONDARY OUTCOMES:
Visual Analog Scale | 8 weeks
  The Visual Analog Scale (VAS) will be used to measure pain intensity by having participants mark their perceived level of pain on a 10-centimeter line ranging from 'no pain' to 'worst pain imaginable.
Scoliosis Research Society-22 (SRS-22) Quality of Life Questionnaire | 8 weeks
  The Scoliosis Research Society-22 (SRS-22) Quality of Life Questionnaire measures the impact of scoliosis on patients' quality of life across five domains: function, pain, self-image, mental health, and satisfaction, using a total of 22 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Eyuboglu, PhD., Study Director — Uskudar University; Mert Ilhan, MSc., Principal Investigator — Uskudar University
Locations (1):
- Uskudar University Physiotherapy and Rehabilitation Application and Research Center, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No